CLINICAL TRIAL: NCT02256033
Title: Effect of Mild Hepatic Impairment (Child-Pugh Class A) on the Single-dose Pharmacokinetics of Istradefylline
Brief Title: Effect of Mild Hepatic Impairment on the Pharmacokinetics of Istradefylline
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Collaborators: Kyowa Hakko Kirin Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 6002-016
Record Dates: First submitted 2014-09-16; First posted 2014-10-03 (Estimated); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Hepatic Impairment
Keywords: Mild hepatic impairment; Healthy volunteer; Istradefylline
MeSH Terms: interventions — istradefylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Istradefylline (Experimental): One 40-mg tablet of istradefylline administered on Day 1.
  Interventions: Drug: Istradefylline

INTERVENTIONS:
Drug: Istradefylline — One 40 mg-tablet administered on Day 1
  Other Names: KW-6002

SUMMARY:
The purpose of this study is to test whether mild liver impairment affects blood levels of istradefylline in humans. Decreased liver function could possibly increase istradefylline levels.

DETAILED DESCRIPTION:
This is a multicenter, open-label, parallel group, single-dose study to determine the single-dose PK of istradefylline in subjects with mild hepatic impairment (HI) (Child-Pugh Class A) and in subjects with normal hepatic function. Ten subjects with mild HI (Child-Pugh Class A) and 10 subjects with normal hepatic function (matched for age, gender, race, and BMI) will be enrolled. Enrollment of the subjects with normal hepatic function will be subsequent to the HI subjects.

ELIGIBILITY:
Inclusion Criteria:

All subjects:

* Non-smoking males and females 18-75 years of age, inclusive;
* Men and women with procreative potential must practice medically reliable double barrier methods of birth control;
* Body mass index (BMI): 18.0-35.0 kg/m2, inclusive:
* Must abstain from drugs and nutrients known as moderate to potent inhibitors/inducers of CYP3A4 and CYP1A enzymes. These agents should be discontinued at least 4 weeks before the istradefylline dose (Day 1) until the Follow-up visit.
* Negative results at Screening and Baseline for the following screening laboratory tests: urine drug screen (amphetamines, barbiturates, benzodiazepines, opiates, cannabinoids, and cocaine). Documented prescription use in subjects with mild HI for medications included in the urine drug of abuse test is permitted as long as the dose is stable for at least 2 weeks;

Subjects with Normal Hepatic Function only

* Medical history without clinically significant or ongoing pathology, which in the opinion of the Investigator will preclude the subject's participation in, or influence the outcome of the study;

Subjects with Mild Hepatic Impairment only

* Stable, mild liver disease (Child-Pugh A [5 to 6 points]); of cryptogenic, post-hepatic, hepatitis B/C virus, or alcoholic origin;
* Stable hepatic impairment, defined as no clinically significant change in disease status within the last 30 days, as documented by the subject's recent medical history;

Additional inclusion criteria apply

Exclusion Criteria:

* Female subjects who are taking oral contraceptives or long-term injectable or implantable hormonal contraceptives, pregnant, lactating, or breast-feeding;
* Known history of treatment for drug or alcohol addiction within the previous 12 months or > 14 untis of alcohol consumption per week, or alcohol consumption within 1 week prior to dosing;
* Positive test results for human immunodeficiency virus (HIV), or Hepatitis B surface antigen;
* Difficulty fasting or eating the standard meals that will be provided;
* Use of tobacco or nicotine-containing products within 90 days of the study start to the Follow-up visit (to be confirmed by urine cotinine test);

Subjects with Hepatic Impairment only

* Severe ascites at Screening;
* History of or current severe hepatic encephalopathy (Grade 3 or higher)
* Any of the following laboratory parameters at screening:

  1. Serum ALT > 5 × the upper limit of normal range (ULN);
  2. Serum albumin < 2.4 g/dL;
  3. Platelet count < 80,000/mm3;
  4. Hemoglobin < 11 g/dL;
  5. Absolute neutrophil count (ANC) < 1.5 × 109/L (< 1.5 × 103/μL);
* Biliary liver cirrhosis or other causes of HI not related to parenchymal disorder and/or disease of the liver, including hepatocellular carcinoma.

Additional exclusion criteria apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Comparison of pharmacokinetic parameter istradefylline (Area under the concentration-time curve [AUC]) between subjects with hepatic impairment and healthy subjects with normal hepatic function using an analysis of variance model | Intermittently for a total of 36 days
  Single-dose pharmacokinetics (PK) of istradefylline in subjects with mild hepatic impairment (HI) (Child-Pugh Class A) and in subjects with normal hepatic function

SECONDARY OUTCOMES:
Number of adverse events and serious adverse events | Continuously for 36 days
  Safety and tolerability will be assessed through review of recorded adverse events and serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Cantillon, M.D., Study Chair — Kyowa Hakko Kirin Pharma, Inc.; Amy Zhang, PhD., Study Director — Kyowa Hakko Kirin Pharma, Inc.
Locations (2):
- United States (2):
  - Orlando Clinical Research Center, Orlando, Florida
  - Noccr/Vrg, Knoxville, Tennessee